CLINICAL TRIAL: NCT02933437
Title: An Observational Study Into the Variety of Electrocardiographic Responses to an Ajmaline Provocation in a Healthy Subjects. What Are the Genetic and Structural Variations Dictating This Response ?
Brief Title: The Response To Ajmaline Provocation in Healthy Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16.0012; 2016-004277-41 (EudraCT Number)
Record Dates: First submitted 2016-08-31; First posted 2016-10-14 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Brugada Syndrome; Sudden Death
Keywords: Brugada syndrome; SCN5A; SCN10A; Ajmaline
MeSH Terms: conditions — Brugada Syndrome; Death, Sudden | interventions — Ajmaline; Prajmaline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Once screened by the investigators, the participants will undergo ajmaline provocation, cardiac magnetic resonance imaging and genotype evaluation
  Interventions: Drug: Ajmaline

INTERVENTIONS:
Drug: Ajmaline — Ajmaline 1milligram/kilogram max dose as bolus intravenous over 10 minutes with continuous ECG monitoring
  Other Names: GILURYTMAL

SUMMARY:
Standard, high lead and sodium channel provoked electrocardiograms of a healthy volunteers will be performed to observe the various ECG changes. Participants will the undergo detailed imaging with cardiac magnetic resonance imaging and deep genotyping to identify structural or genetic variants which might dictate the electrocardiographic patterns at rest and with sodium channel provocation.

DETAILED DESCRIPTION:
The investigators will recruit healthy subjects without a history of cardiac symptoms or a family history of sudden death or premature arrhythmogenic cardiac disease. Participants will undergo electrocardiographic phenotype assessment with standard and high lead electrocardiogram and sodium channel provocation. Detailed cardiac structural examination will be performed with cardiac magnetic resonance imaging to look for any variation in mainly right ventricular outflow tract structure and myocardial architecture. Participants will also undergo targeted genomic sequencing to look for variations in genes encoding for cardiac sodium channel.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic healthy Volunteers

Exclusion Criteria:

* • Any prior cardiovascular illness

  * Previous cardiac symptoms.
  * History of unexplained syncope
  * Any family history of proven sudden cardiac death or unexplained sudden death either in adulthood or infancy.
  * Those unable to provide a two generation family history
  * Abnormal resting ECG
  * Any contraindications to cardiac magnetic resonance imaging
  * Pregnant or breastfeeding women
  * Intercurrent use of any medication known to be contraindicated in Brugada Syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-22 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The qualitative and quantitative effects of ajmaline provocation on parameters of cardiac conduction in healthy subjects using the surface electrocardiogram | ten minutes
  The investigators will be undertaking quantitative analysis of the changes in cardiac conduction observed in the presence of ajmaline. This is measured in time intervals in milliseconds (ms) and magnitude of electrical conduction which will be expressed in millivolts (mv), but can also be expressed in millimetres (mm). The investigators will use the latter to quantify area changes which will be expressed as millimetres squared (mm2). A quantitive description of the electrocardiographic patterns observed will also be performed in addition to further qualitative analysis of vectors created by the variety of ECG morphologies observed, this geometrical assessment will be measured in degrees. As this is a cohort of healthy volunteers the variations observed are anticipated to be part of the "normal" variation, therefore the statistical analysis of these findings will be as a cohort not individual.

SECONDARY OUTCOMES:
The influence of normal variations in right ventricular outflow tract dimensions on the electrocardiographic response to ajmaline provocation in healthy subjects using cardiac magnetic resonance imaging. | intraoperative
  Using existing cardiac magnetic resonance imaging modality, cardiac dimensions will be measured in millimetres (mm). This includes wall thickness and internal cavity size. Additionally volumetric assessment for chamber size will be made using millilitres (ml), this allows for a 3 dimensional appreciation. Using contrast agents, an assessment of the composition of cardiac muscle can be made and can identify the presence or absence of "myocardial fibrosis,"as a binary outcome measure. Further methods will be used to quantify the degree of fibrosis if observed, this will be expressed as a percentage (%) area of fibrosis divided by total area of myocardium multiplied by 100. The location of this fibrosis within the heart will also be noted.
Genotype linkage analysis of the electrocardiographic response to ajmaline provocation in healthy subjects using candidate gene and gene wide association studies. | through study completion, an average of 2 years
  Targeted genetic sequencing of the sodium channel genes SCN5A and SCN10A and gene wide association studies for rare variations

CONTACTS AND LOCATIONS:
Overall Officials: Elijah Behr, MD, Principal Investigator — St George's, University of London
Locations (1):
- St George's University Of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No